CLINICAL TRIAL: NCT02738710
Title: Comparison of Post-operative Pain at Umbilical Wound After Laparoscopic Cholecystectomy With Transumbilical Versus Infraumbilical Incision
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thammasat University (Other)
Responsible Party: Principal Investigator, Boonying Siribumrungwong, Dr., Thammasat University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MTU-EC-SU-1-042/59
Record Dates: First submitted 2016-04-05; First posted 2016-04-14 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Pain, Postoperative; Gallstone
MeSH Terms: conditions — Pain, Postoperative; Gallstones

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- transumbilical wound (Experimental): transumbilical incision
  Interventions: Procedure: transumbilical incision
- infra umbilical wound (Active Comparator): infra umbilical incision
  Interventions: Procedure: Infra umbilical incision

INTERVENTIONS:
Procedure: transumbilical incision — incision within umbilicus
  Arms: transumbilical wound
Procedure: Infra umbilical incision — incision about 1 cm below umbilicus
  Arms: infra umbilical wound

SUMMARY:
This study compare outcomes (i.e. pain, wound infection, and patient satisfaction) between infra-umbilical vs. trans-umbilical incision after Laparoscopic cholecystectomy

DETAILED DESCRIPTION:
Infra-umbilical wound have been used for a while with aim at improving cosmoses of the incision. Formerly, standard incision for laparoscopic cholecystectomy was infra-umbilical wound. However, no study directly compare these types of incisions in term of postoperative pain, wound infection, and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* elective laparoscopic cholecystectomy
* willing to participate

Exclusion Criteria:

* pregnancy
* immunocompromised host
* on continuous ambulatory peritoneal dialysis
* morbid obesity (Body mass index > 35 kg/m2)
* End-stage renal disease with hemodialysis dependent
* ascites
* uncontrolled coagulopathy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2016-09; Primary Completion 2017-09 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | 7 days postoperatively
  visual analog scale (0-10)

SECONDARY OUTCOMES:
wound infection | at 1 week and 1 month postoperatively
  yes or no according to Center for Disease Control and Prevention (CDC) criteria
patient satisfaction | 1 week and 3 months postoperatively
  Visual analog scale (0-10)

CONTACTS AND LOCATIONS:
Overall Officials: Trilak Chunsurisap, Study Chair — Thammasat University Hospital
Locations (1):
- Thammasat University Hospital, Khlong Luang, Pathumtani, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Siribumrungwong B, Chunsirisub T, Limpavitayaporn P, Tongyoo A, Sriussadaporn E, Mingmalairak C, Thowprasert W, Thakkinstian A. Comparison of postoperative pain at umbilical wound after conventional laparoscopic cholecystectomy between transumbilical and infraumbilical incisions: a randomized control trial. Surg Endosc. 2019 May;33(5):1578-1584. doi: 10.1007/s00464-018-6447-y. Epub 2018 Oct 22. PMID 30350096